CLINICAL TRIAL: NCT02967354
Title: [11C]5-Hydroxy-tryptophan Positron Emission Tomography for Assessment of Islet Mass During Progression of Type 2 Diabetes
Brief Title: [11C]5-Hydroxy-tryptophan PET for Assessment of Islet Mass in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Per-Ola Carlsson (Other)
Responsible Party: Sponsor-Investigator, Per-Ola Carlsson, Professor, Senior consultant, Uppsala University Hospital
Organization: Uppsala University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Dnr 2012/302
Record Dates: First submitted 2016-11-08; First posted 2016-11-18 (Estimated); Results first posted 2017-11-29 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Type2 Diabetes
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Healthy control (Experimental): Healthy control
  Interventions: Radiation: Positron emission tomography with the tracer [11C]5-hydroxy-tryptophan
- Obese with oral antidiabetic drugs (Experimental): BMI>30, Type 2 diabetes treated with oral antidiabetic drugs
  Interventions: Radiation: Positron emission tomography with the tracer [11C]5-hydroxy-tryptophan
- Obese, treated with oral antidiabetic drugs + insulin (Experimental): BMI>30, Type 2 diabetes treated with oral antidiabetic drugs + insulin
  Interventions: Radiation: Positron emission tomography with the tracer [11C]5-hydroxy-tryptophan
- Normal weight, treated with oral antidiabetic drugs (Experimental): BMI 20-26. Type 2 diabetes treated with oral antidiabetic drugs
  Interventions: Radiation: Positron emission tomography with the tracer [11C]5-hydroxy-tryptophan
- Normal weight, treated with oral antidiabetic drugs + insulin (Experimental): BMI 20-26. Type 2 diabetes treated with oral antidiabetic drugs + insulin
  Interventions: Radiation: Positron emission tomography with the tracer [11C]5-hydroxy-tryptophan

INTERVENTIONS:
Radiation: Positron emission tomography with the tracer [11C]5-hydroxy-tryptophan — Estimation of islet mass by PET using the tracer [11C]5-hydroxy-tryptophan

SUMMARY:
Cross-sectional study to investigate subjects at different stages of type 2 diabetes development with expected stratification of pancreatic islet mass. Non-diabetic individuals were assigned as control. The primary outcome was the [11C]5-hydroxy-tryptophan uptake and retention in the pancreas as a surrogate marker for the endogenous islet mass.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes fulfilling criteria for the four different study groups, or healthy volunteers

Exclusion Criteria:

* Ongoing pregnancy
* Renal failure (GFR<60 ml/min)
* Magnetic metal parts in the body
* Ongoing treatment with selective serotonin receptor inhibitors

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-01; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

REFERENCES:
- [Derived] Carlbom L, Espes D, Lubberink M, Martinell M, Johansson L, Ahlstrom H, Carlsson PO, Korsgren O, Eriksson O. [11C]5-hydroxy-tryptophan PET for Assessment of Islet Mass During Progression of Type 2 Diabetes. Diabetes. 2017 May;66(5):1286-1292. doi: 10.2337/db16-1449. Epub 2017 Feb 28. PMID 28246291

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy Control | Obese With Oral Antidiabetic Drugs | Obese, Treated With Oral Antidiabetic Drugs + Insulin | Normal Weight, Treated With Oral Antidiabetic Drugs | Normal Weight, Treated With Oral Antidiabetic Drugs + Insulin
Started | 8 | 7 | 9 | 7 | 8
Completed | 8 | 7 | 9 | 7 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Control | Obese With Oral Antidiabetic Drugs | Obese, Treated With Oral Antidiabetic Drugs + Insulin | Normal Weight, Treated With Oral Antidiabetic Drugs | Normal Weight, Treated With Oral Antidiabetic Drugs + Insulin | Total
Number analyzed (Participants) | 8 | 7 | 9 | 7 | 8 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (6.2) | 56.7 (10.1) | 61.8 (7.2) | 60.3 (10.8) | 66.3 (5.4) | 61.8 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 2 | 2 | 4 | 14
  Male | 4 | 5 | 7 | 5 | 4 | 25
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 8 | 7 | 9 | 7 | 8 | 39
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 28.1 (3.4) | 33.3 (2.6) | 33.2 (3.6) | 25.1 (2.4) | 25.8 (1.4) | 29.2 (2.7)

OUTCOME MEASURES:

1. Primary Outcome: [11C]5-hydroxy-tryptophan Uptake in the Pancreas
Description: Uptake of tracer with correlation to functional measurement with glucose-potentiated arginine stimulation of insulin release
Time Frame: Within two weeks after functional measurement with glucose potentiated arginine stimulation of insulin release
Population: Two healthy controls and two individuals in the group "Normal weight, treated with oral antidiabetic drugs + insulin were not included in the analysis because of not being able to participate in the PET scan, pancreatic anatomical abnormality or insufficient image quality.
Measure: Mean (Standard Deviation); unit: % of injected dose
Arm/Group | Healthy Control | Obese With Oral Antidiabetic Drugs | Obese, Treated With Oral Antidiabetic Drugs + Insulin | Normal Weight, Treated With Oral Antidiabetic Drugs | Normal Weight, Treated With Oral Antidiabetic Drugs + Insulin
Number analyzed (Participants) | 6 | 7 | 9 | 7 | 6
% of injected dose | 0.17 (0.04) | 0.21 (0.10) | 0.20 (0.07) | 0.23 (0.11) | 0.15 (0.14)
Statistical Analysis 1: Comparison: Healthy Control vs Obese With Oral Antidiabetic Drugs vs Obese, Treated With Oral Antidiabetic Drugs + Insulin vs Normal Weight, Treated With Oral Antidiabetic Drugs vs Normal Weight, Treated With Oral Antidiabetic Drugs + Insulin; Test type: Superiority; p = 0.5875, ANOVA — Treshold for significance P<0.05

2. Secondary Outcome: Pancreatic Perfusion
Description: Uptake of radioactive water with correlation to functional measurement with glucose-potentiated arginine stimulation of insulin release
Time Frame: Within two weeks after functional measurement with glucose potentiated arginine stimulation of insulin release
Population: Some individuals in the study population were not included in the analysis because of not being able to participate in the PET scan, pancreatic anatomical abnormality or insufficient image quality.
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Healthy Control | Obese With Oral Antidiabetic Drugs | Obese, Treated With Oral Antidiabetic Drugs + Insulin | Normal Weight, Treated With Oral Antidiabetic Drugs | Normal Weight, Treated With Oral Antidiabetic Drugs + Insulin
Number analyzed (Participants) | 6 | 6 | 8 | 7 | 6
ml/min | 84.37 (18.17) | 134.90 (47.84) | 107.72 (32.91) | 72.20 (18.88) | 59.82 (51.16)
Statistical Analysis 1: Comparison: Healthy Control vs Obese With Oral Antidiabetic Drugs vs Obese, Treated With Oral Antidiabetic Drugs + Insulin vs Normal Weight, Treated With Oral Antidiabetic Drugs + Insulin; Test type: Superiority; p = 0.0065, ANOVA — Treshold for significance P<0.05

3. Secondary Outcome: Pancreatic Volume
Time Frame: Within two weeks after functional measurement with glucose potentiated arginine stimulation of insulin release
Population: Some participants were not included in the analysis because of not being able to participate in the imaging, pancreatic anatomical abnormality or insufficient image quality.
Measure: Mean (Standard Deviation); unit: cm^3
Arm/Group | Healthy Control | Obese With Oral Antidiabetic Drugs | Obese, Treated With Oral Antidiabetic Drugs + Insulin | Normal Weight, Treated With Oral Antidiabetic Drugs | Normal Weight, Treated With Oral Antidiabetic Drugs + Insulin
Number analyzed (Participants) | 6 | 6 | 8 | 7 | 6
cm^3 | 67.68 (8.90) | 88.54 (23.99) | 98.96 (23.85) | 64.1 (13.46) | 53.39 (41.17)
Statistical Analysis 1: Comparison: Healthy Control vs Obese With Oral Antidiabetic Drugs vs Obese, Treated With Oral Antidiabetic Drugs + Insulin vs Normal Weight, Treated With Oral Antidiabetic Drugs vs Normal Weight, Treated With Oral Antidiabetic Drugs + Insulin; Test type: Superiority; p = 0.0072, ANOVA — Treshold for significance P<0.05

4. Secondary Outcome: Pancreatic Fat Content
Time Frame: Within two weeks after functional measurement with glucose potentiated arginine stimulation of insulin release
Population: Some of the study participants were not included in the analysis because of not being able to participate in the MRI scan, pancreatic anatomical abnormality or insufficient image quality.
Measure: Mean (Standard Deviation); unit: % of pancreatic volume
Arm/Group | Healthy Control | Obese With Oral Antidiabetic Drugs | Obese, Treated With Oral Antidiabetic Drugs + Insulin | Normal Weight, Treated With Oral Antidiabetic Drugs | Normal Weight, Treated With Oral Antidiabetic Drugs + Insulin
Number analyzed (Participants) | 7 | 6 | 8 | 7 | 6
% of pancreatic volume | 11.33 (7.62) | 11.54 (10.30) | 8.75 (2.97) | 9.58 (9.37) | 9.72 (7.97)
Statistical Analysis 1: Comparison: Healthy Control vs Obese With Oral Antidiabetic Drugs vs Obese, Treated With Oral Antidiabetic Drugs + Insulin vs Normal Weight, Treated With Oral Antidiabetic Drugs vs Normal Weight, Treated With Oral Antidiabetic Drugs + Insulin; Test type: Superiority; p = 0.9472, ANOVA — Treshold for significance P<0.05

5. Secondary Outcome: Hepatic Fat Content
Time Frame: Within two weeks after functional measurement with glucose potentiated arginine stimulation of insulin release
Population: Some of the study participants were not included in the analysis because of not being able to participate in the MRI scan or insufficient image quality.
Measure: Mean (Standard Deviation); unit: % of liver volume
Arm/Group | Healthy Control | Obese With Oral Antidiabetic Drugs | Obese, Treated With Oral Antidiabetic Drugs + Insulin | Normal Weight, Treated With Oral Antidiabetic Drugs | Normal Weight, Treated With Oral Antidiabetic Drugs + Insulin
Number analyzed (Participants) | 7 | 6 | 8 | 6 | 6
% of liver volume | 5.30 (3.15) | 14.40 (7.18) | 13.42 (7.14) | 5.50 (2.98) | 9.01 (4.55)
Statistical Analysis 1: Comparison: Healthy Control vs Obese With Oral Antidiabetic Drugs vs Obese, Treated With Oral Antidiabetic Drugs + Insulin vs Normal Weight, Treated With Oral Antidiabetic Drugs vs Normal Weight, Treated With Oral Antidiabetic Drugs + Insulin; Test type: Superiority; p = 0.0048, ANOVA — Treshold for significance P<0.05

ADVERSE EVENTS:
Arm/Group | Healthy Control | Obese With Oral Antidiabetic Drugs | Obese, Treated With Oral Antidiabetic Drugs + Insulin | Normal Weight, Treated With Oral Antidiabetic Drugs | Normal Weight, Treated With Oral Antidiabetic Drugs + Insulin
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7 | 0/9 | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7 | 0/9 | 0/7 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No